CLINICAL TRIAL: NCT00437788
Title: The Effect of a Digital Photograph of the Patient in a CT Scan Examination on the Quality of Diagnosis by the Radiologist
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: 1907CTIL
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-01

CONDITIONS: Healthy
Keywords: imaging

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Whenever a scan is accessed through the PACS system a scanned document or digital picture may be displayed automatically. In this study the technician will take a digital picture of the patient who will be undergoing the CT scan. This way the radiologist will be able to view the patient's face before viewing the scan.

The hypothesis is that viewing a digital picture of the patient before viewing the CT scan will improve the quality of diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient who are to be scanned by ct

Exclusion Criteria:

* Disabled

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000

CONTACTS AND LOCATIONS:
Overall Officials: yonatan turner, MD, Principal Investigator — Shaheed Ziaur Rahman Medical College